CLINICAL TRIAL: NCT05851794
Title: Intraoperative Endomanometric Laparoscopic Nissen Fundoplication Improves Postoperative Outcomes in Large Sliding Hiatus Hernia With Severe Gastroesophageal Reflux Disease (DeMeester Score >100). A Retrospective Comparative Study.
Brief Title: Intraoperative Endomanometric Laparoscopic Nissen Fundoplication Improves Postoperative Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, professour of general and laparoscopic surgery, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GERD
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endomanometric laparoscopic Nissen fundoplication (Active Comparator): use endomanometry and endoscope during laparoscopic Nissen fundoplication
  Interventions: Procedure: endomanometric guided LNF
- laparoscopic Nissen fundoplication alone (Active Comparator): laparoscopic Nissen fundoplication only
  Interventions: Procedure: laparoscopic Nissen fundoplication alone

INTERVENTIONS:
Procedure: endomanometric guided LNF — use of endomanometry during LNF
  Arms: endomanometric laparoscopic Nissen fundoplication
Procedure: laparoscopic Nissen fundoplication alone — laparoscopic Nissen fundoplication alone
  Arms: laparoscopic Nissen fundoplication alone

SUMMARY:
Laparoscopic Nissen fundoplication (LNF) is a surgical intervention for gastroesophageal reflux disease (GERD); however, it can be followed by recurrent symptoms or complications that may affect patient satisfaction. Intraoperative endomanometric evaluation of esophagogastric competence and pressure, combined with LNF in patients with large sliding hiatus hernia (>5cm) with severe GERD (DeMeester score >100), is needed.This is a retrospective, multicenter, comparative study. Baseline characteristics, initial reflux symptoms, preoperative and postoperative antacid medication use, postoperative complications (dysphagia and gas bloat syndrome), recurrent symptoms, and satisfaction were collected from a prospective database. Outcomes measures were recurrent reflux symptoms, postoperative side-effects, and satisfaction with surgery. Quantitative data were compared between the studied groups using the independent t-test or Mann-Whitney U test for normally and non-normally distributed numerical variables, respectively

DETAILED DESCRIPTION:
Laparoscopic Nissen fundoplication (LNF) is a surgical intervention for gastroesophageal reflux disease (GERD); however, it can be followed by recurrent symptoms or complications that may affect patient satisfaction. Intraoperative endomanometric evaluation of esophagogastric competence and pressure, combined with LNF in patients with large sliding hiatus hernia (>5cm) with severe GERD (DeMeester score >100), is needed.

Study design: This is a retrospective, multicenter, comparative study. Baseline characteristics, initial reflux symptoms, preoperative and postoperative antacid medication use, postoperative complications (dysphagia and gas bloat syndrome), recurrent symptoms, and satisfaction were collected from a prospective database. Outcomes measures were recurrent reflux symptoms, postoperative side-effects, and satisfaction with surgery. Quantitative data were compared between the studied groups using the independent t-test or Mann-Whitney U test for normally and non-normally distributed numerical variables, respectively.

This study contributes to the mounting evidence for the effectiveness of endomanometric use during LNF. Intraoperative HRM and Endoscope were feasible in all patients and demonstrated that the clinical outcomes for endomanometric NF were favorable from an effectiveness and safety standpoint.

ELIGIBILITY:
Inclusion Criteria:

* patients 18≥ years with large sliding hiatus hernia (> 5 cm) with severe GERD patients (DeMeester score >100)with typical symptoms and successful medical management (due to quality of life considerations, life-long need medication intake or cost) or patients with unresponsive or inadequate symptom control despite eight weeks of adequate medical therapy with or without extra-esophageal Atypical symptoms that are related to GERD(cough, Globus, or hoarseness) confirmed diagnosis by hypotensive lower esophageal sphincter confirmed by HRM and a positive pH/impedance test (based on DeMeester scores)
* fitness and consenting for surgery
* patients that completed three year follow up period,
* with esophagitis

Exclusion Criteria:

* <18years,
* pregnancy,
* Patients unfit for surgery [ comorbid condition like severe cardiac illness, chronic respiratory diseases, chronic renal failure, and bleeding disorder],
* Non cooperative or lost patients for regular follow up,
* Patients who had undergone previous antireflux surgery or who required a concurrent abdominal procedure at the same time as fundoplication (eg, cholecystectomy), -
* psychiatric disorders.
* esophageal dysmotility,

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
DeMeester score (0-3) | 3 years
  0 is best while 3 is worst
dysphagia score(0-3) | 3 years
  0 is best while 3 is worst

IPD SHARING:
Plan to Share IPD: No